CLINICAL TRIAL: NCT06107517
Title: DREAMS-OT Trial: Delirium Reduction Through Early Activation in Motivating and Sleep Promoting Routines: A Randomized Controlled Trial of Occupational Therapy for ICU Patients After Coronary Artery Bypass Graft (CABG) Surgery
Acronym: DREAMS-OT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other); National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022/00936
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-08

CONDITIONS: Delirium, Postoperative
Keywords: Delirium; Coronary Artery Bypass Grafting; Occupational Therapy; Intensive Care Units; Randomized Controlled Trial
MeSH Terms: conditions — Emergence Delirium; Delirium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DREAMS-OT Arm (Intervention Group) (Experimental): Patients will receive an early and intensive occupational therapy protocol starting within the first 15 hours after extubation.
  Interventions: Other: DREAMS-OT
- Standard Care Arm (Control Group) (No Intervention): Standard care OT as per current ICU setting

INTERVENTIONS:
Other: DREAMS-OT — Patients will receive the DREAMS-OT protocol 3 times per day, 20 minutes per therapy session.
  Intervention frequency will be confirmed with a feasibility trial. If not feasible to maintain 3 times per day, the intervention will still be maintained at the same intensity of 1 hour per day, with a graded approach.
  Arms: DREAMS-OT Arm (Intervention Group)

SUMMARY:
The goal of this randomized controlled trial (RCT) is to compare the effectiveness of the DREAMS-OT intervention with standard care in reducing post-Coronary Artery Bypass Graft (CABG) delirium in patients undergoing CABG.

The aims of the study are:

* Conduct a prospective randomized controlled trial comparing the effectiveness of the DREAMS-OT intervention with standard care in reducing post-CABG delirium in Cardiothoracic Intensive Care Unit (CTICU)
* To conduct a nested cost-effectiveness study

The study team will compare intervention group and standard care group (control group) to see if there is a reduction in the incidence of delirium in patients 5 days post-CABG.

ELIGIBILITY:
Inclusion Criteria:

* Patients deemed medically suitable for elective CABG surgery
* Patients aged 21 years and above
* Patients who are English or Mandarin speaking.
* Patients who are able to provide consent

Exclusion Criteria:

* Patients who speak other languages are excluded due to the language requirements of certain outcome measures.
* Patients with premorbid severe hearing impairment, severe cognitive impairment, progressive neurological disorders and psychological disorders will be excluded.
* Patients with surgical complications resulting in profuse bleeding from any invasive sites, septic shock unresponsive to maximal treatment, and those who are moribund or have an expected mortality within 48 hours will be excluded.
* Pregnant women will also be excluded from the study as well.
* Patients who develop delirium before initiation of the treatment are also excluded from the study.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Delirium | Day 1 of post-CABG (AM and PM), Day 2 of post-CABG (AM and PM), Day 3 of post-CABG (AM and PM), Day 4 of post-CABG (AM and PM), Day 5 of post-CABG (AM and PM); (+/- 1 day for last measurement)
  Incidence of delirium within 5 days of undergoing CABG. Measured using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) assessment tool

SECONDARY OUTCOMES:
Length of Stay | 3-months post-CABG (+/- 1 month)
  Length of stay in ICU and hospital in days
Duration of Delirium | Day 1 of post-CABG (AM and PM), Day 2 of post-CABG (AM and PM), Day 3 of post-CABG (AM and PM), Day 4 of post-CABG (AM and PM), Day 5 of post-CABG (AM and PM)
  Duration of delirium in subgroup of participants who develop delirium
Sleep Quality | 2 weeks prior to operation (Baseline measurement, +/- 2 weeks), Day 3 of post-CABG, Day 4 of post-CABG (+/- 1 day), 3 months post-CABG for 3 consecutive days (+/- 1 month)
  Sleep quality (Duration of Total Sleep, Light Sleep, Deep Sleep and Rapid Eye Movement (REM) Sleep in hours) as measured with Oura Ring, a wearable sleep tracking device
Functional Status | Day 5 of post-CABG (+/- 1 day)
  Function status using Acute Care Index of Function (ACIF)
Physical Status | Day 5 of post-CABG (+/- 1 day), 3 months post-CABG (+/- 1 month)
  Physical status measurement using Functional Independence Measure (FIM)
Cognitive status | 2 weeks prior to operation (Baseline measurement, +/- 2 weeks), Day 5 of post-CABG (+/- 1 day), 3 months post-CABG (+/- 1 month)
  Cognitive status measurement using Montreal Cognitive Assessment (MoCA)
Psychological State | 2 weeks prior to operation (Baseline measurement, +/- 2 weeks), Day 5 of post-CABG (+/-1 day), 3 months post-CABG (+/- 1 month)
  Psychological state using the Hospital Anxiety and Depression Scale (HADS)
Cognitive status | 3-months post-CABG (+/- 1 month)
  Weekly Calendar Planning Activity (WCPA)

OTHER OUTCOMES:
Richmond Agitation Sedation Scale (RASS) | Day 1 of post-CABG (AM and PM), Day 2 of post-CABG (AM and PM), Day 3 of post-CABG (AM and PM), Day 4 of post-CABG (AM and PM), Day 5 of post-CABG (AM and PM)
  RASS which will be used for CAM-ICU assessment (primary outcome measure).
European System for Cardiac Operative Risk Evaluation (EuroSCORE) 2 | 3-months post-CABG (+/- 1 month)
  EuroSCORE 2 is used to assess the risk of heart surgery of participants before their CABG surgery
Charlson Comobility Index (CCI) | 3-months post-CABG (+/- 1 month)
  Predicts mortality for participant before CABG surgery
Clinical Frailty Index (CFI) | 3-months post-CABG (+/- 1 month)
  Measure health status of participant before surgery
ICU Mobility Score | Day 1 of post-CABG, Day 3 of post-CABG, Day 4 of post-CABG (+/- 1 day, or until day of ICU discharge)
  Measure ICU mobility during ICU stay
Pain Score | Day 1 of post-CABG, Day 2 of post-CABG, Day 3 of post-CABG, Day 4 of post-CABG, Day 5 of post-CABG (+/- 1 day, or until day of ICU discharge)
  Measure pain score of participant
Time on Mechanical Ventilation and Ventilator Free Days | 3-months post-CABG (+/- 1 month)
  Time on Mechanical Ventilation of participant in hours and Ventilator Free Days in days during ICU stay
30-day readmission and mortality | 3-months post-CABG (+/- 1 month)
  Incidence of readmission or death within 30 days after CABG
Short Form (36) Health Survey (SF-36) | 2 weeks prior to operation (Baseline measurement, +/- 2 weeks), 3-months post-CABG (+/- 1 month)
  Measure quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Su Ren Wong, Principal Investigator — National University Hospital, Singapore